CLINICAL TRIAL: NCT04992494
Title: Treatment for Migraine and Mood (Team-M): A Pilot Trial of a Mindfulness-based Training Program
Brief Title: Treatment for Migraine and Mood (Team-M)
Acronym: TEAM-M
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01911; R01AT011005 (NIH)
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Migraine; Depression
MeSH Terms: conditions — Migraine Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) (Experimental): Mindfulness-based cognitive therapy delivered by Telephone
  Interventions: Behavioral: MBCT-Telephone
- MBCT-V (Mindfulness-Based Cognitive Therapy - Video) (Experimental): Mindfulness-based cognitive therapy delivered by Video
  Interventions: Behavioral: MBCT-Video

INTERVENTIONS:
Behavioral: MBCT-Telephone — Mindfulness-based cognitive therapy (MBCT) comprised of 8 weekly classes delivered via telephone by a licensed clinical psychologist certified to teach MBCT, following treatment fidelity guidelines from NIH's Behavioral Change Consortium.
  The program involves a commitment of 1 hour per week for 8 weeks. During the sessions, subjects will learn cognitive and mindfulness skills to help manage and cope with depression. Each weekly session consists of: check-in, instruction, skill building, discussion, and a home-based practice assignment.
  Arms: MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone)
Behavioral: MBCT-Video — Mindfulness-based cognitive therapy (MBCT) comprised of 8 weekly classes delivered via WebEx video-conferencing by a licensed clinical psychologist certified to teach MBCT, following treatment fidelity guidelines from NIH's Behavioral Change Consortium.
  The program involves a commitment of 1 hour per week for 8 weeks. During the sessions, subjects will learn cognitive and mindfulness skills to help manage and cope with depression. Each weekly session consists of: check-in, instruction, skill building, discussion, and a home-based practice assignment.
  Arms: MBCT-V (Mindfulness-Based Cognitive Therapy - Video)

SUMMARY:
The researchers propose a two-arm pilot study of telephone and video delivered Mindfulness-based Cognitive Therapy (MBCT-T and MBCT-V) in people with migraine and depressive symptoms.

DETAILED DESCRIPTION:
This study aims to set the stage for a future definitive large-scale Phase III trial in patients with migraine and depressive symptoms. This first phase is aimed at fidelity optimization of MBCT-T and MBCT-V in people with migraine (defined by the International Classification of Headache Disorders - 3) and depressive symptoms (defined by empirical cut-offs on the Patient Health Questionnaire - 9).

ELIGIBILITY:
Inclusion Criteria:

* Currently meets ICHD-3 criteria for migraine using the Structured Diagnostic Interview for Headache
* Self-reported 4-14 headache days per month, with at least one attack meeting migraine criteria
* Score between 5-14 on the PHQ-9
* Age ≥ 18
* Ability to read and speak English
* Capacity to consent

Exclusion Criteria:

* Meeting ICHD-3 criteria for persistent headache attributed to traumatic injury to the head (post-traumatic headache) on the Structure Diagnostic Interview for Headache
* Changes in preventive migraine medication or anti-depressant medication within 6 weeks of intake; changes in longer-term migraine prevention (onobotulinum toxin A, anti-calcitonin gene related peptide treatment) within 3 months of intake
* Comorbid psychiatric illness or clinical features that would interfere with participant's ability to participate in or receive benefit from the MBCT intervention, including but not limited to: active suicidal ideation; recent history of psychosis or mania; borderline, histrionic or narcissistic personality disorder; cognitive impairment; sensory disabilities
* Prior history of engaging in formal mindfulness-based interventions including: MBSR, MBCT, Acceptance and Commitment therapy, Dialectical Behavior Therapy
* Current meditation practice >3x/week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Shallcross, ND, MPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone): Mindfulness-based cognitive therapy delivered by Telephone
  MBCT-Telephone: Mindfulness-based cognitive therapy (MBCT) comprised of 8 weekly classes delivered via telephone by a licensed clinical psychologist certified to teach MBCT, following treatment fidelity guidelines from NIH's Behavioral Change Consortium.
  The program involves a commitment of 1 hour per week for 8 weeks. During the sessions, subjects will learn cognitive and mindfulness skills to help manage and cope with depression. Each weekly session consists of: check-in, instruction, skill building, discussion, and a home-based practice assignment.
- MBCT-V (Mindfulness-Based Cognitive Therapy - Video): Mindfulness-based cognitive therapy delivered by Video
  MBCT-Video: Mindfulness-based cognitive therapy (MBCT) comprised of 8 weekly classes delivered via WebEx video-conferencing by a licensed clinical psychologist certified to teach MBCT, following treatment fidelity guidelines from NIH's Behavioral Change Consortium.
  The program involves a commitment of 1 hour per week for 8 weeks. During the sessions, subjects will learn cognitive and mindfulness skills to help manage and cope with depression. Each weekly session consists of: check-in, instruction, skill building, discussion, and a home-based practice assignment.
Period: Overall Study
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video)
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13) | 44 (14) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 7 | 13
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Treatment Session Adherence Rate
Description: Treatment Session Adherence is a measure of treatment feasibility and is defined as the number of scheduled treatments that were attended by the participants. This measure will be assessed through electronic monitoring of the attendance logs of each treatment session. A treatment arm will be considered feasible if participants attended/read 75% of sessions on average.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: Number of sessions attended
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video)
Number analyzed (Participants) | 8 | 8
Number of sessions attended | 7.88 (0.35) | 8 (0)

2. Primary Outcome: Average Client Satisfaction Questionnaire Score (CSQ-8)
Description: The CSQ-8 is an 8-item generic standardized self-report tool to measure satisfaction with health and human services received by individuals and families. An overall score is calculated by summing the respondent's rating (item rating) score for each scale item. For the CSQ-8 version, scores range from 8 to 32, with higher values indicating higher satisfaction. A threshold score of greater than or equal to 24 is the cut-off for "Acceptability."
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video)
Number analyzed (Participants) | 8 | 7
score on a scale | 29.3 (3.2) | 28.3 (3.7)

3. Primary Outcome: Mean Score on MBCT-T/V Adherence & Competence Scales (MBCT-TACS)
Description: The mindfulness-based cognitive therapy (MBCT)-TACS is an assessment of treatment fidelity in terms of adherence and competence. The scores per session are recorded between 0-3 and averaged to get the total score. The total range of score is 0-3; the higher the score, the higher the fidelity.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video)
Number analyzed (Participants) | 8 | 8
score on a scale | 2.9 (0.3) | 2.8 (0.4)

4. Primary Outcome: Homework Assignment Completion Rate
Description: Defined as the proportion of assigned home-based practice that participants completed each week.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: proportion of assignments completed
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video)
Number analyzed (Participants) | 6 | 8
proportion of assignments completed | 0.77 (0.15) | 0.57 (0.21)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events were systematically assessed using weekly questionnaires during the study intervention. Serious adverse events and all-cause mortality were not monitored/assessed.
Arm/Group | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/8 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MBCT-T (Mindfulness-Based Cognitive Therapy - Telephone) (N=8) | MBCT-V (Mindfulness-Based Cognitive Therapy - Video) (N=6)
Increased severity of migraine (Nervous system disorders) | 1 | 0
Flashback (General disorders) | 2 | 1
COVID infection (Infections and infestations) | 2 | 2
Worsening hyperthyroidism (Endocrine disorders) | 1 | 0
Worsening mood (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04992494/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04992494/ICF_000.pdf